CLINICAL TRIAL: NCT07072767
Title: Increasing Live Donor Kidney Transplantation Through Video-based Education and Mobile Communication
Brief Title: Hybrid Dissemination Study of A Digital-Analog Intervention to Increase Live Donor Kidney Transplantation
Acronym: KIDNEYTIME+
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Liise Kayler, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00014971
Record Dates: First submitted 2025-01-31; First posted 2025-07-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: End-Stage Renal Disease; Chronic Kidney Diseases; Kidney Transplant; Living Kidney Donor
Keywords: pilot randomized trial; behavioral intervention
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KidneyTime-2 with human support (Experimental): KidneyTIME-2 is a multicomponent mobile education-outreach intervention to increase patient- and network-to-donor self-learning and outreach, about living donor kidney transplantation. Human guide support offered over a 6 month period to encourage use of the intervention and donor outreach.
  Interventions: Behavioral: Digital education outreach intervention for kidney transplant access and human guide
- KidneyTime-2 without human support (Active Comparator): KidneyTime-2 is a multicomponent mobile education-outreach intervention to increase patient- and network-to-donor self-learning and outreach, about living donor kidney transplantation. Routine clinical support from non-study sources through usual Transplant Center protocols including clinic provider communications.
  Interventions: Behavioral: Digital education outreach intervention for kidney transplant access only (unguided)

INTERVENTIONS:
Behavioral: Digital education outreach intervention for kidney transplant access and human guide — Receives (1) donor search materials, (2) electronic resource access messages, (3) practical assistance to use the intervention and empower taking the outreach action and (4) telephonic human guide
  Arms: KidneyTime-2 with human support
Behavioral: Digital education outreach intervention for kidney transplant access only (unguided) — Receives (1) donor search materials, (2) electronic resource access messages, and (3) practical assistance to use the intervention and empower taking the outreach action.
  Arms: KidneyTime-2 without human support

SUMMARY:
The study is a 2-arm randomized controlled trial among patients referred for kidney transplant evaluation at a single transplant center to compare the effects of a digital-analog intervention to increase living-donor kidney transplant access (KidneyTIME+) with or without human guide . Following consent and baseline assessment, participants are randomized, stratified by self-reported race, with equal allocation to 2 treatment arms: the KidneyTIME+ intervention with or without human guide.

DETAILED DESCRIPTION:
Over a 3-year period the investigators will conduct a pilot 2-arm parallel randomized trial among patients referred for kidney transplantation at a single transplant center to compare the effects of KidneyTIME+ with or without ongoing human support for KTX access over 6 months of intervention use and follow-up.

Participants will be recruited from the Transplant program at Erie County Medical Center, a safety-net hospital in Buffalo, New York. Each week, electronic records will be accessed to identify patients and their carers who present for transplant evaluation at the transplant center for a kidney transplant, are aged 18 years and older, speak English, and are competent to provide informed consent . The investigators will exclude patients previously exposed to any component of the intervention, listed for transplantation at another center, and seeking multiorgan transplantation.

A stakeholder Advisory Council, whose members include patients and care partners, will review and provide ongoing feedback on the recruitment and retention plan. They will also provide input on assistive dissemination tools for organizations to engage individuals to use the resource.

Each potential participant will be invited to the study by a researcher who will describe the study and answer and questions, and provide a copy of the consent form describing study procedures and potential risks.

Those who sign electronic consent to participate will be asked to complete a baseline sociodemographic and pre-test survey. Upon completion, computer-generated randomization will stratify participants by self-reported race (Black versus Other), with equal allocation to 2 treatment arms: the KidneyTIME+ intervention with or without human guide. Condition assignment of each participant will be concealed from transplant providers, but participants will become aware of their treatment assignment once they access the human guide.

KidneyTIME+ is a digital-analog intervention with human support. It is based on animated video education targeted to patients, donors, and support persons, designed to address knowledge gaps and concerns about kidney transplantation and living donation that were identified in literature reviews, formative research, and video development studies as critical for optimal prospective kidney recipient and donor participation in LDKT. Other key components include (1) personalized donor outreach materials, (2) email reminders about study resources, and (3) practical assistance to ensure access to intervention, advise use the intervention and encourage outreach actions. All components of the intervention were developed through a user-centered design approach by involving kidney failure patients and social network members, to improve usability and increase the likelihood of uptake.

In both intervention and control arms, the investigators chose 6 videos from the entire series to be delivered sequentially for a total duration of 13 minutes. The video content sets the stage for the intervention and introduces the viewer to an overview of LDKT, including addressing common misconceptions about live kidney donation, donor eligibility, donor evaluation, kidney paired donation, donation costs, and donor recovery. After completing the proscribed videos everyone then receives weekly emails with links to the full video curriculum centralized on a website and other local resources. Email messages introduce study videos and features and local resources that may interest users, provide access links, and encourage video viewing and sharing. Messages will be personalized with the participants name and provide researchers contact information. The videos on the website are activated for sharing through various modalities, including text, email, Facebook, and Twitter. The website also contains templates and examples for other donor outreach materials and practical engagement materials to promote awareness of the website. The website is open access from any electronic device. Finally, at clinic appointments participants will receive practical assistance to use intervention materials.

In the intervention arm, donor outreach will be supported by telephonic human guides who will provide tailored implementation support in 7 areas that include ensuring access, advising use, recommending features, encouraging donor outreach, and referrals to clinical services, support groups, community resources. Human guides will interact with participants over a 6-month period.

Control participants will not receive human guide support.

All participants routinely receive educational materials from non-study sources through usual Transplant Center protocols including written materials and clinical provider communications. Providers may recommend the study website or individuals may find it on their own.

After completing the proscribed video education, all participants will be invited to fill out serial surveys at 6 months post-evaluation. Participants will receive up to 6 reminders (5 automatic and 1 personalized) to complete surveys. At study conclusion, participants may be invited to an exit interview.

ELIGIBILITY:
Inclusion Criteria:

* referred to the transplant center for a kidney transplant
* aged 18 years and older
* speaks English

Exclusion Criteria:

* Previously exposed to any component of the intervention
* Listed for a kidney transplant at another center (multilisted)
* Seeking multiorgan transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Living donor inquiry | Baseline, post baseline 6 months
  Count of living donor inquires to the transplant center on behalf of the study participants within 6 months from enrollment. Each inquiry (telephone call, email, letter) is counted and added to a discrete field for all patients in the electronic medical record.

SECONDARY OUTCOMES:
LDKT Perceived understanding | Baseline, post baseline 6 months
  Developed specifically for this study as a measure of perceived understanding about LDKT as delivered in the intervention condition. In this 4 item 4-point Likert questionnaire, total scores range from 4-16 with higher scores indicating greater LDKT-related understanding. The scale captures different dimensions of understanding including kidney transplant navigation, awareness of services, and donor outreach.
LDKT Conversational self-efficacy | Baseline, post baseline 6 months
  A 2-item survey testing confidence to communicate about LDKT with others. Items are rated on a scale of 1 to 4, total scores range from 2-8. Higher scores indicate greater confidence to communicate about LDKT with others.
LDKT Beliefs scale | Baseline, post baseline 6 months
  Developed specifically for this study as a measure of patients' beliefs about LDKT. Questions were drawn from existing measures in the literature. We created a 2-item scale. One item captured the degree to which a person believes that LDKT is an advantage. The other item assessed the degree to which a person believes their social network is healthy enough to donate a kidney. Items are rated on a scale of 1 to 4. Total scores range from 2-8 with higher scores indicate greater concerns about live kidney donation.
Donor outreach behaviors | Baseline, post baseline 6 months
  A measure of ongoing outreach toward living donor kidney transplantation. To assess LDKT action behaviors patients will be asked whether they had done any of 14 related behaviors adapted from existing measures in the literature. Patients who indicated they had done the action will be counted and scores will range from 0 to 14. Higher scores indicate more outreach.

OTHER OUTCOMES:
Time to waiting-list placement | 12 months
  The first time from evaluation to active placement on the kidney transplant waiting list will be assessed via medical record review.
Intervention Acceptability | Post-baseline 6 months
  16-item survey assessing intervention usage, ease of use, and usefulness. Each question has 4 Likert-scale options bounded by strongly agree and strongly disagree or multiple responses specific to the question. Total scores range from 16-64 with higher scores indicate greater intervention acceptability.
Patient perception of donor offer | Baseline, post baseline 6 months
  A one item question asking participants if someone has agreed to donate a kidney to them, with the options of answering 'yes', 'no', or 'maybe'.

CONTACTS AND LOCATIONS:
Locations (1):
- Erie County Medical Center, 462 Grider Street, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
No funding available for sharing